CLINICAL TRIAL: NCT01809145
Title: Testing Hypersensitivity to Metals in Sarcoidosis Patients With Occupational Exposure, Using the MELISA Test.
Brief Title: Testing Hypersensitivity to Metals in Sarcoidosis Patients by Applying the MELISA Test.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-13-LF-0683-CTIL
Record Dates: First submitted 2013-03-07; First posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; occupational exposure; MELISA
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- metal hypersensitivity (Other): peripheral blood test for metal hypersensitivity (MELISA test)
  Interventions: Other: MELISA test

INTERVENTIONS:
Other: MELISA test — MELISA test for hypersensitivity to metals in sarcoidosis

SUMMARY:
The purpose of this study is to apply the MELISA test, that diagnose hypersensitivity to metals, in Sarcoidosis patients with occupational exposure.

DETAILED DESCRIPTION:
Peripheral blood from sarcoidosis patients with occupational anamnesis that involves exposure to metals will be sent to MELISA Medica in Stockholm Sweden. The MELISA test will examine hypersensitivity to metals that can be related to the granulomatous response of sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

Biopsy confirmed sarcoidosis Granulomatous disease Occupational anamnesis with exposure to metals

Exclusion Criteria:

Patients with interstitial disease No occupational anamnesis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
MELISA test | 30 days
  Using the MELISA test in peripheral blood, in order to find hypersensitivity to metals that can be related to the granulomatous response of sarcoidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Fireman, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel, Israel